CLINICAL TRIAL: NCT00206336
Title: An Open-label Study to Determine the Efficacy and Safety of Topiramate in the Treatment of Tourette Syndrome (CAPSS-286)
Brief Title: An Open-label Study to Determine the Efficacy and Safety of Topiramate in the Treatment of Tourette Syndrome.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Principal Investigator, Joseph Jankovic, Principal Investigator, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAPSS-286
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Tourette Syndrome
MeSH Terms: conditions — Tourette Syndrome | interventions — Topiramate; Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- topiramate (Experimental): Topiramate open label
  Interventions: Drug: Topiramate (drug)

INTERVENTIONS:
Drug: Topiramate (drug) — Topiramate 25 mg to 200 mg
  Other Names: Topamax

SUMMARY:
Previous studies using topiramate in Tourette subjects have shown that with the use of this medication subjects report that their tics get better. The purpose of this study is to study if topiramate improves the symptoms of Tourette syndrome, such as motor tics, or other associated symptoms such as attention or obsessive-compulsive problems.

DETAILED DESCRIPTION:
In order to enroll in this study, you must have completed the Double-Blind phase of CAPSS-176 or discontinued the Double-Blind phase of CAPSS-176 after a minimum of 6 weeks because it has been determined that your symptoms of Tourette Syndrome were getting worse. You must also continue to meet the specific inclusion and exclusion criteria outlined in CAPSS-176.

The Titration/Maintenance Period: will last for 10 weeks, as it did during CAPSS-176. During the Titration and Maintenance Periods of the study, you will visit the study center 4 times. Visit 1 (Day 1) will be the same day as your final visit for CAPSS-176. You will have had a physical examination (including sitting blood pressure, pulse and weight), a urine pregnancy test if you are a female that is capable of having a child and been given the scale that measures the severity of your symptoms of Tourette Syndrome as part of the final visit procedures for CAPSS-176. This information will also be included as part of Visit 1.

During this visit, a blood sample will be taken (approximately 3 teaspoons) and tested to rule out any abnormalities and to make sure that your liver is working properly and your electrolytes are normal. You will also be asked to answer questions for the scale that measures your symptoms, if any, of attention deficit hyperactivity disorder (A-D/HD). If you have Bipolar II Disorder, you will be asked to answer questions for one scale that measures your symptoms of mania. If you have obsessive-compulsive disorder (OCD), you will be asked to answer questions for one scale that measures those symptoms. The study doctor or his staff will complete two scales that assess the severity of your condition.

If you continue to be eligible for the study, you will begin the Titration Period of the study by taking 1 tablet of commercial topiramate 25 mg in the evening. This will be Day 1 of the study. After one week of this phase of the study, your topiramate dose will be increased to 2 tablets of topiramate (50 mg total), one tablet in the morning and one in the evening. Your topiramate dose may continue to be increased until you have reached the dose level the study doctor determines to be appropriate for you, or, you are taking a maximum dose of 200 mgs per day of topiramate. Your study doctor may adjust your topiramate dose as necessary.

During the study, you will be expected to visit your study doctor or his staff again on Day 28 (Visit 2), Day 56 (Visit 3) and Day 70 (Visit 4) after beginning treatment. Extra visits may be scheduled at the discretion of your study doctor. At each visit, you will have your blood pressure, pulse and weight measured. You will be asked how you are feeling and if you have started taking any new medications or had changes in other medications you may be taking. All of the scales that were completed at Visit 1, and the scale that was completed at the final visit of CAPSS-176, will be completed again at each visit. You will have a urine pregnancy test performed at each visit if you are a female capable of having a child. The test must be negative to continue in the study. You will have blood drawn again (approximately three teaspoons) at Visits 2 and 4 to make sure that your liver is functioning properly and your electrolytes are normal.

You will be called between Visits 1 and 2 (Day 14 of the study) and Visits 2 and 3 (Day 42 of the study) on the telephone by one of the people working on this study. During these phone calls you will be asked how you are feeling, if you have had any changes in medications you are taking and how you are doing with topiramate.

Commercial topiramate will be provided in 25 mg tablets.Study medication is provided in child resistant bottles.All bottles should be returned(regardless of whether they are partial, empty or full) at each visit. It is important that you follow your study doctor or his staff's instructions on when and how to take the topiramate. At Visit 4 (Day 70), you will be given instructions about reducing your topiramate dose gradually for the next week. You will visit the study doctor or his staff again on Day 77 (Visit 5) after you have completely stopped taking the topiramate.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must continue to meet the specific inclusion criteria outlined in either CAPSS-176 or CAPSS-198 to enroll in this protocol.
* Subjects must have completed the Double-Blind Phase or discontinued the Double-Blind Phase after a minimum of 6 weeks due to lack of efficacy (defined by a CGI improvement score of >6 [much worse or very much worse]) in either CAPSS-176 or CAPSS-198.
* Subjects or their parents/guardians, must be able to read and comprehend written instructions and willing to complete all scales and assessments required by this protocol.
* After full explanation of the study, subjects, or their parent/legally authorized representatives, must demonstrate their willingness to participate by signing an informed consent form. If applicable, pediatric subjects capable of giving assent must sign the assent form.
* Subjects must continue their current treatment for tics, treatment of comorbid symptoms or treatment of A-D/HD at the dose level established prior to entry in the Double-Blind Phase of CAPSS-176 or CAPSS-198.

Exclusion Criteria:

* Subjects must continue to meet the specific exclusion criteria outlined in either CAPSS-176 or CAPSS-198 to enroll in this protocol.
* Subjects who have SGOT and/or SGPT levels greater than 2 times the upper limit of the normal range from the last visit in either CAPSS-176 or CAPSS-198 will not be permitted to enroll in the current study.

Ages: 7 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Jankovic, MD, Principal Investigator — Baylor College of Medicine

REFERENCES:
- [Background] Jankovic J, Jimenez-Shahed J, Brown LW. A randomised, double-blind, placebo-controlled study of topiramate in the treatment of Tourette syndrome. J Neurol Neurosurg Psychiatry. 2010 Jan;81(1):70-3. doi: 10.1136/jnnp.2009.185348. Epub 2009 Sep 1. PMID 19726418

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Topiramate
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Topiramate
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.5 (9.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in TTS
Description: A component of the Yale Global Tic Severity Scale (YGTSS), the change from baseline in Total Tic Score (TTS) at visit 5 (day 70) is the pre-defined primary endpoint. The Total Tic Score is a summation of the Total Motor Tic and Total Phonic Tic Scores. The Overall Impairment Rating is rated on a 50-point scale anchored by 0 (No impairment) and 50 (Severe impairment).
Time Frame: baseline to Day 70
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Topiramate
Number analyzed (Participants) | 20
units on a scale | -14.29 (10.47)

ADVERSE EVENTS:
Arm/Group | Topiramate
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 4/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topiramate (N=20)
headache (General disorders) | 3 (3)
cognitive slowing (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Because of the small sample size and open label design we decided not to pursue publication of the extension study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No